CLINICAL TRIAL: NCT02184286
Title: An Investigation of the Potential Pharmacokinetic Interaction Between Nevirapine (VIRAMUNE®) and Saquinavir-sgc (Fortovase®) in HIV-1 Infected Patients
Brief Title: Pharmacokinetic Interaction Between Nevirapine and Saquinavir-sgc in HIV-1 Infected Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1100.1280
Record Dates: First submitted 2014-07-08; First posted 2014-07-09 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine

ARMS (1):
- Nevirapine + Saquinavir-sgc (Experimental)
  Interventions: Drug: Nevirapine; Drug: Saquinavir-sgc

INTERVENTIONS:
Drug: Nevirapine — 200 mg q.d. days 1-14 followed by 200 mg b.i.d. days 15-28
Drug: Saquinavir-sgc — 1600 mg b.i.d. from pre trial to day 28

SUMMARY:
The objectives of this study are to determine the effects of nevirapine on the steady-state pharmacokinetics of saquinavir-sgc and to determine the effects of saquinavir-sgc on the steady-state pharmacokinetics of nevirapine. This study will also evaluate the pharmacokinetics of nevirapine in combination with saquinavir-sgc compared to historical controls treated with nevirapine but without saquinavir-sgc.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between the ages of 18 and 65 years who are seropositive for HIV-1 antibody by an ELISA test and confirmed by an alternative method, e.g. Western blot
* Patients who meet the following laboratory parameters:

  * Granulocyte count ≥ 1000 cells/mm3
  * Hemoglobin ≥ 9.0 g(dL (men and women)
  * Platelet count ≥ 75,000 cells/mm3
  * Alkaline phosphatase ≤ 3.0 times the upper limit of normal
  * Serum glutamic oxalo-acetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) ≤ 3.0 times the upper limit of normal
  * Total bilirubin ≤ 1.5 times the upper limit of normal
* Patients receiving a stable antiretroviral regimen, including saquinavir-sgc (Fortovase®) 1600 mg b.i.d. in the 28 days prior to visit 1
* Female patients of childbearing potential must be willing to use a reliable form of contraception, which should include a medically approved form of barrier contraception
* Patients able to provide written informed consent and comply with study requirements
* Patients with a viral load less than 400 copies/mL

Exclusion Criteria:

* Female patients who are pregnant or breastfeeding
* Patients requiring systemic treatment with corticosteroids or drugs known to be hepatic enzyme inducers or inhibitors in the 14 days prior to visit 1. Such substances in these categories include macrolide antibiotics (erythromycin, clarithromycin, azithromycin, dirithromycin), azole antifungals (ketoconazole, fluconazole, itraconazole), rifampin, rifabutin, and phenytoin
* Patients with previous exposure to (or are currently being treated with) non-nucleoside reverse transcriptase inhibitors (NNRTIs)
* Patients receiving a protease inhibitor other than saquinavir-sgc (Fortovase®) in the 28 days prior to visit 1
* Patients receiving any investigational drug, antineoplastic agent or radiotherapy other than local skin radiotherapy treatment in the 12 weeks prior to visit 1
* Patients with malabsorption, severe chronic diarrhea or patients unable to maintain adequate oral intake
* Patients with a current history of intravenous drug abuse, alcohol or substance abuse (within the last year)
* Patients undergoing treatment for an active infection
* Patients who are heavy smokers (≥ 20 cigarettes or cigars per day)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 1999-05; Primary Completion 2000-02 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | up to 12 hours post-dose on days 1 and 28
Time of maximum concentration (Tmax) | up to 12 hours post-dose on days 1 and 28
Minimum observed concentration (Cmin) | up to 12 hours post-dose on days 1 and 28
Area under the plasma concentration time profile over the steady-state dosing interval (AUCτ) | up to 12 hours post-dose on days 1 and 28
Systemic clearance (Cl/F) | up to 12 hours post-dose on days 1 and 28

SECONDARY OUTCOMES:
Change in HIV RNA levels | Baseline and day 28
Change in cluster differentiation 4 positive (CD4+) count | Baseline and day 28
Number of patients with adverse events | up to 28 days